CLINICAL TRIAL: NCT02747485
Title: Impact of Diffuse Myocardial Fibrosis on the Ventricular Function in Regurgitant Left-Sided Valve Heart Diseases " The DIFFUsE Study "
Brief Title: Impact of Diffuse Myocardial Fibrosis on the Ventricular Function in Regurgitant Left-Sided Valve Heart Diseases ( The DIFFUsE Study)
Acronym: DIFFUsE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2016-11; 2015-A00587-42 (Other: ansm)
Record Dates: First submitted 2016-04-19; First posted 2016-04-21 (Estimated); Last update posted 2019-03-07 (Actual); Status verified 2019-03

CONDITIONS: Valve Heart Diseases
MeSH Terms: conditions — Heart Valve Diseases | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- organic left-sided regurgitant valve (Experimental)
  Interventions: Device: Cardiac MRI; Biological: blood samples; Procedure: myocardial biopsy; Genetic: blood samples

INTERVENTIONS:
Device: Cardiac MRI
Biological: blood samples — Serum levels of biomarkers of myocardial fibrosis (galectine-3 and ST2) will be measured
Procedure: myocardial biopsy
Genetic: blood samples — extract DNA to look for genomic mutations associated with the disease.

SUMMARY:
New strategies are needed to early detect myocardial involvement in these diseases. Histological studies showed that diffuse fibrosis and cardiomyocyte hypertrophy precede the LV remodelling (dilatation) observed by cardiac imaging. Quantification of LV diffuse myocardial fibrosis using magnetic resonance imaging (MRI) could reach this goal. Recently, contrast enhanced cardiac MRI has been used to measure the extracellular volume fraction (ECV) of the myocardium, and it has been able to detect diffuse myocardial fibrosis. In diseases in which increased collagen deposition enlarges the extra-cellular space, the ECV can act as a fibrosis index. ECV is correlated with the amount of fibrosis measured by histology. Left ventricular overloads induced by regurgitant VHD result in cardiomyocyte hypertrophy and diffuse fibrosis. Other methods can be used to estimate the degree of myocardial fibrosis such as the serum level of galectine-3 or ST2. Moreover, although the pathophysiological mechanisms leading to the occurrence of myocardial fibrosis differ in patients with various cardiac diseases, the cellular effectors of fibrotic remodelling are common and involve similar signalling pathways. At the cellular level, key progression of ventricular hypertrophy is associated with increased cardiomyocytes apoptosis and fibrosis, suggesting that these two processes are responsible for the transition.

To our knowledge, no study has analysed the impact of the rate of myocardial diffuse fibrosis, non-invasively estimated by ECV, in the risk of LV dysfunction during MR and AR, especially after surgery. The measurement of ECV could become an important tool for risk stratification in left-sided regurgitant VHD. Thus, it would provide an early marker of LV myocardial involvement before the occurrence of global remodeling, might help physicians in surgical decision, and would improve prognosis. This is an innovative original project because it uses modern imaging modalities to answer to a crucial question. The clinical implications would be important because this work would modify the international surgical indications of MR and AR in order to finally improve the prognosis of patients with this frequent heart disease. Moreover, investigators will analyze the genetic factors that can influence the myocardial reaction resulting from these regurgitations, which will improve the quality of this work and offer new future perspectives.

Investigators hypothesize that the ECV measurement could be used as an early predictor of LV dysfunction in the left-sided valve regurgitations.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive patients referred for organic MR and/or AR at least moderate to severe according to the ESC guidelines criteria⁴ will be eligible. The moderate to severe criteria will defined by echocardiography as followed:
* MR: an effective regurgitant orifice area (EOA) >30mm2 and/or a regurgitant volume (RV) >45mL
* AR: an EOA >20mm2 and/or a RV >45mL

Exclusion Criteria:

* Age < 18 years
* Pregnancy
* Impossibility to maintain a decubitus position
* Arrhythmia that do not allow an ECG synchronization during MRI
* Hemodynamic instability
* Indication of urgent surgery
* Known coronary artery disease
* Severe arterial hypertension
* Cardiomyopathy
* Claustrophobia
* Gadolinium intolerance
* Implantable medical devices that do allow to perform MRI
* Severe renal insufficiency with clearance <35 mL/min
* Vulnerable patients
* Acute infective endocarditis
* Aortic dissection
* Moderate or severe mitral stenosis (mitral area <1.5cm2/m2)
* Moderate or severe aortic stenosis (aortic area <0.8cm2/m2, or Vmax>3m/s, or mean gradient>30mmHg)
* Previous cardiac surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 316 (Estimated)
Dates: Start 2016-05 (Actual); Primary Completion 2020-08 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
the rate of diffuse myocardial fibrosis | 6 months

SECONDARY OUTCOMES:
Correlations between ECV and the global longitudinal strain and the serum level of Galectin-3 and ST2 | 42 months
Correlations between ECV changes and genetic factors | 42 months
correlations between ECV and the severity of the regurgitation | 42 months
correlation between ECV and the myocardial deformation quantified by speckle tracking echocardiography (2D Strain) | 42 months

CONTACTS AND LOCATIONS:
Overall Officials: Catherine GEINDRE, Study Director — Assistance Publique Hopitaux De Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, Bouche DU Rhone, France

IPD SHARING:
Plan to Share IPD: Undecided